CLINICAL TRIAL: NCT06624670
Title: A Multi-centre, Randomised, Placebo-controlled, Double-blind, Parallel-group Trial to Evaluate Safety and Efficacy of Spesolimab (BI 655130) in Adult Patients With Ulcerative Pyoderma Gangrenosum (PG) Who Require Systemic Therapy
Brief Title: A Study to Test Whether Spesolimab Helps People With a Skin Condition Called Pyoderma Gangrenosum
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1368-0140; 2024-514306-31-00 (Registry Identifier: CTIS (EU)); U1111-1306-8055 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2024-09-30; First posted 2024-10-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pyoderma Gangrenosum
MeSH Terms: conditions — Pyoderma Gangrenosum | interventions — spesolimab; Prednisone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Spesolimab (Experimental)
  Interventions: Drug: Spesolimab; Drug: Prednisone; Drug: Prednisolone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo matching to spesolimab; Drug: Prednisone; Drug: Prednisolone

INTERVENTIONS:
Drug: Spesolimab — Solution for infusion
  Arms: Spesolimab
Drug: Placebo matching to spesolimab — Placebo matching to spesolimab
  Arms: Placebo
Drug: Prednisone — Prednisone
Drug: Prednisolone — Prednisolone

SUMMARY:
The purpose of this study is to find out whether a medicine called spesolimab helps people with pyoderma gangrenosum (PG). The main aim is to see whether spesolimab leads to closure of PG ulcers. This study is open to adults with ulcerative PG with at least 1 ulcer that measures between 5 cm^2 to 80 cm^2 in size.

This study has 2 parts. In Part 1, participants are put into groups randomly, which means by chance. 1 group gets spesolimab and the other group gets placebo. Placebo infusions look like spesolimab infusions, but do not contain any medicine. Every participant has a 2 in 3 chance of getting spesolimab. For the first 8 weeks, participants also take corticosteroid medicine by mouth.

In Part 2, participants are put into groups again. Participants without open ulcers have an equal chance of getting spesolimab or placebo. Participants with open skin ulcers will get spesolimab.

In both parts, participants receive spesolimab or placebo as an infusion into a vein every 4 weeks.

Participants are in the study for about 1.5 years. During this time, they visit the study site 20 times. At study visits, doctors check the participant's skin for signs of PG. The doctors also regularly check participants' health and take note of any unwanted effects. The results of the groups are compared to see whether the treatment works.

ELIGIBILITY:
Inclusion criteria:

1. Adult trial participants, aged ≥18 years (if local legislation for age of consent differs, then local legislation will be followed) at screening.
2. Signed and dated written informed consent in accordance with International Council on Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
3. A confirmed diagnosis of ulcerative pyoderma gangrenosum (PG) (≥10 points on the PARACELSUS score) that requires systemic therapy in the opinion of the investigator. The diagnosis needs to be confirmed by an Adjudication Committee. Trial participants with mixed PG subtypes are eligible as long as the target lesion is of the ulcerative subtype.
4. At least one measurable (defined as measuring ≥5 cm^2) PG ulcer. In trial participants with more than one PG ulcer, the target PG ulcer will be selected by the investigator and confirmed by external Adjudication Committee.
5. At the time of the Screening Visit, a maximum duration of 6 months since the target ulcer in the current PG episode was diagnosed. Target ulcers >6 months since diagnosis are allowed if they are active and progressing, as judged by the investigator and confirmed by an Adjudication Committee.
6. Women of childbearing potential (WOCBP) must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria and instructions on the duration of use is provided in the participant information and in the protocol.

Exclusion criteria:

1. Trial participants with non-PG lesions.
2. Trial participants with a target PG ulcer measuring >80 cm^2.
3. Trial participants with chronic, non-inflamed PG wounds or ulcers that are not responsive to immunosuppressive therapy, as determined by an Adjudication Committee.
4. Presence of active ulcer infection at the Screening Visit (unless treated and resolved prior to administration of the first dose of trial medication) based on investigator assessment.
5. Presence of persistent or recurring bacterial infection requiring systemic antibiotic therapy; or clinically significant viral, fungal, or parasitic infections within 2 weeks prior to the Screening Visit. Any such infection must be resolved, with treatment completed ≥2 weeks prior to the Screening Visit. No new/recurrent infections should have occurred prior to Visit 2.
6. "Active or latent tuberculosis (TB)

   * Participants with active TB are excluded
   * Participants with latent TB may be included if treatment of latent TB, as per local guidelines, is initiated prior to randomization and completed during the course of the trial."
7. Chronic or acute infections including Human immunodeficiency virus (HIV) infections and viral hepatitis (including occult hepatitis); the corresponding laboratory tests will be performed during screening. A trial participant can be re-screened if the trial participant was treated and is cured from the acute infection.
8. Severe, progressive, or uncontrolled hepatic disease, defined as >3x Upper Limit of Normal (ULN) elevation in Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) or alkaline phosphatase, or >2x ULN elevation in total bilirubin.

Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-02-04 (Actual); Primary Completion 2027-04-12 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
Achievement of complete closure (PGAR-100 (100% pyoderma gangrenosum area reduction)) of the target PG ulcer at any time up to Week 26 and confirmed at the next consecutive visit (at least 2 weeks later) | Up to Week 28.
  PGAR-100 is defined as complete closure and re-epithelisation of a PG ulcer without drainage and requirements for dressing.

SECONDARY OUTCOMES:
Key secondary endpoint: Achievement of PGAR-100 of the target PG ulcer at Week 26 confirmed at the next consecutive visit (at least 2 weeks later) | Up to Week 28.
  PGAR-100 is defined as complete closure and re-epithelisation of a PG ulcer without drainage and requirements for dressing.
Achievement of 50% area reduction (PGAR-50) of the target PG ulcer at any time up to Week 26 | Up to Week 26.
  Achievement of a PGAR-50 defines an area reduction of a PG ulcer from baseline by 50%.
Achievement of ≥ 3 point reduction in NRS Pain score from baseline at Week 26 | At baseline and at Week 26.
  Numeric Rating Scale for Pain (NRS Pain) is a unidimensional measure of pain intensity. It is a 11-point numeric scale, in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of their pain, with 0 representing "no pain" and 10 representing "worst pain imaginable". Trial participant is asked to report their pain intensity in the last 24 h.
Achievement of a DLQI of ≤ 5 at Week 26 | At Week 26.
  Dermatology Life Quality Index (DLQI) is a trial participant-administered, quality of life questionnaire consisting of 10 questions that cover 6 domains (symptoms and feelings, daily activities, leisure, work and school, personal relationships, problems with treatment).
  Response categories include "not relevant" or "not at all" (score of 0), "a little" (score of 1), "a lot" (score of 2) and "very much" (score of 3). Question 7 is a "yes"/ "no" question where "yes" is scored as 3. DLQI total score is calculated by summing the scores of each question, resulting in a range of 0 to 30, with higher scores indicating more impairment of a trial participant's quality of life.
Achievement of complete response | At Week 26.
  Complete response (CR), defined as all ulcers completely closed and re- epithelised without drainage and requirements for dressing, as assessed by the investigator).
Achievement of PGAR-100 of any measurable PG ulcer (≥5 cm^2 at baseline) at any time up to Week 26 and confirmed at the next consecutive visit (at least 2 weeks later) | Up to Week 28.
  PGAR-100 is defined as complete closure and re-epithelisation of a PG ulcer without drainage and requirements for dressing.
Achievement of PGAR-100 of all measurable PG ulcers (≥5 cm^2 at baseline) at any time up to Week 26 and confirmed at the next consecutive visit (at least 2 weeks later) | Up to Week 28.
  PGAR-100 is defined as complete closure and re-epithelisation of a PG ulcer without drainage and requirements for dressing.
Time to recurrence among trial participants who had achieved CR at Week 26 up to Week 52 | Up to Week 52.
  Recurrence is defined as emergence of the disease (PG ulcer[s]) at the previous ulcer sites(s) or emergence of any new PG ulcer(s).

CONTACTS AND LOCATIONS:
Locations (90):
- United States (19):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Medical Dermatology Specialists Phoenix, Phoenix, Arizona
  - University of California Irvine, Irvine, California
  - University of Miami, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Dawes Fretzin Clinical Research Group, LLC-Indianapolis -68995, Indianapolis, Indiana
  - Tulane University Hospital and Clinic, New Orleans, Louisiana
  - Brigham and Women's Hospital, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Dartmouth Hitchcock Clinics Heater Road, Lebanon, New Hampshire
  - Dermatology at Lake Success, Lake Success, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Red River Research Partners, LLC, Fargo, North Dakota
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health and Sciences University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Epiphany Dermatology, Lewisville, Texas
  - University of Utah Health, Murray, Utah
- Argentina (3):
  - CIPREC, CABA
  - Hospital Italiano de Buenos Aires, CABA
  - Instituto de Especialidades de la Salud Rosario, Rosario
- Australia (3):
  - Skin and Cancer Foundation, Darlinghurst, New South Wales
  - Royal North Shore Hospital-St Leonards-20807, St Leonards, New South Wales
  - Alfred Hospital, Melbourne, Victoria
- Austria (2):
  - Medical University of Graz State Hospital - University Hospital Graz, Graz
  - LKH Salzburg University Hospital, Salzburg
- UZ Leuven, Leuven, Belgium
- Brazil (2):
  - Chronos Pesquisa Clinica, Brasília
  - Faculdade de Medicina do ABC, Santo André
- Canada (5):
  - Rejuvenation Dermatology Clinic, Edmonton, Alberta
  - University of Alberta Hospital (University of Alberta), Edmonton, Alberta
  - Women's College Hospital, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Centre de Recherche Saint-Louis, Québec
- China (13):
  - Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - The Second Xiangya Hospital Of Central South University, Changsha
  - West China Hospital, Sichuan University, Chengdu
  - The First Affiliated Hospital, Zhejiang University, Hangzhou
  - The Second Affiliated Hospital Zhejiang University School of Medicine, Hangzhou
  - Hangzhou Third People's Hospital, Hangzhou
  - Shandong Provincial Hospital of Dermatology, Jinan
  - Shanghai Skin Disease Hospital, Shanghai
  - The University of Hong Kong-Shenzhen Hospital, Shenzhen
  - Wuhan Union Hospital, Wuhan
  - Second Affiliated Hospital of Xi'an JiaoTong University, Xi'an
- HUS Tulehduskeskus /Ihosairauksien linja, Helsinki, Finland
- France (3):
  - HOP Privé Antony, Antony
  - Hôpital de l'Archet, Nice
  - HOP Saint-Louis, Paris
- Germany (5):
  - Charité - Universitätsmedizin Berlin, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen AöR, Essen
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Würzburg AÖR, Würzburg
- Italy (7):
  - Fondazione IRCCS Ca'Granda-Ospedale Maggiore Policlinico, Milan
  - Azienda Ospedaliera Universitaria Pisana, Pisa
  - Istituti Fisioterapici Ospitalieri, Roma
  - AOU Policlinico Umberto I, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Istituto Clinico Humanitas, Rozzano (MI)
  - Azienda Ospedaliera Universitaria Citta Della Salute E Della Scienza Di Torino, Torino
- Japan (8):
  - Fujita Health University Hospital, Aichi, Toyoake
  - Hokkaido University Hospital, Hokkaido, Sapporo
  - Hyogo College of Medicine Hospital, Hyogo, Nishinomiya
  - Mie University Hospital, Mie, Tsu
  - Tohoku University Hospital, Miyagi, Sendai
  - Jichi Medical University Hospital, Tochigi, Shimotsuke
  - Teikyo University Hospital, Tokyo, Itabashi-ku
  - Nihon University Itabashi Hospital, Tokyo, Itabashi-ku
- Malaysia (3):
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Sarawak General Hospital, Kuching
  - Hospital Pulau Pinang-Pulau Pinang-21953, Pulau Pinang
- Norway (2):
  - Oslo Universitetssykehus HF, Rikshospitalet, Oslo
  - Helse Stavanger, Stavanger Universitetssykehus, Stavanger
- Poland (2):
  - Military Medical Institute- National Research Institute, Warsaw
  - Cityclinic Medical and Psychological Clinic Matusiak Partnership, Wroclaw
- Portugal (4):
  - CHUC - Centro Hospitalar e Universitário de Coimbra, EPE, Coimbra
  - ULS de São José, E.P.E. - Hospital Sto. António Capuchos, Lisbon
  - ULS de Santa Maria, E.P.E, Lisbon
  - ULS de Santo Antônio, E.P.E - Centro Hospitalar Universitário de Santo António, Porto
- Spain (2):
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
- Karolinska Universitetssjukhuset Solna, Stockholm, Sweden
- University Hospital Zurich, Zurich, Switzerland
- Taiwan (3):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chang Gung Medical Foundation (CGMF) - Linkou Bran, Linkou District
  - National Taiwan University Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com